CLINICAL TRIAL: NCT06057844
Title: Molecular Imaging of Active Venous Thrombus With Positron Emission Tomography (PET)
Acronym: THROMPET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 29BRC20.0202
Record Dates: First submitted 2023-09-19; First posted 2023-09-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Venous Thromboembolism (VTE)
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non applicable (Other)
  Interventions: Other: Additional blood sampling

INTERVENTIONS:
Other: Additional blood sampling — Once you have been informed and have given your consent, 2 tubes of venous blood (citrated tubes of approximately 5 milliliters (ml) each) will be taken after the blood donation to enable in vitro thrombus formation. The entire sample will be used, and no surplus will be kept in the bank.

SUMMARY:
Venous thromboembolism (VTE), which includes deep vein thrombosis (DVT) and/or pulmonary embolism (PE), is a major public health issue. VTE is the third most common acute cardiovascular pathology, after myocardial infarction and stroke.

Diagnostic accuracy is essential in the case of VTE, in order to select patients for whom anticoagulant treatment is necessary, and to avoid long-term treatment of patients who will derive no benefit from it.

The management of patients with suspected PE is based on diagnostic strategies that use either ventilation-perfusion planar lung scintigraphy or thoracic angioscanner imaging as the cornerstone. These 2 techniques correspond to what might be termed "negative" imaging, i.e. visualization of the vascular repercussions downstream of an obstruction, whatever its nature.

A research prospect in the field of VTE diagnosis is the direct marking of the various elements of the active venous thrombus, which could correspond to "positive" thrombus imaging.

Numerous studies have already investigated the role of molecular imaging in the diagnosis of VTE, especially in the diagnosis of DVT. However, these studies used conventional scintigraphy to evaluate these tracers, a technique lacking in sensitivity and with insufficient spatial resolution.

Nuclear medicine and molecular imaging have undergone a technological revolution since the early 2000s, with the development of positron emission tomography (PET). The technical advantages of PET over conventional scintigraphy include greater sensitivity and higher spatial resolution (4 mm for PET vs. 12 mm for conventional scintigraphy), which may have been the limiting factor in studies already carried out.

The aim of this project is to develop a new radiopharmaceutical for use in PET scans, a biomarker of active venous thrombus, with a view to improving the diagnosis of MVTE and hence patient management.

ELIGIBILITY:
Inclusion Criteria:

Major patient (≥18 years), voluntary blood donor, with no notable medical history altering coagulation (i.e. known thrombophilia, active cancer), no chronic pathology, no current treatment.

Exclusion Criteria:

Minor patient (<18 years); known chronic pathology; long-term treatment including anti-platelet aggregation therapy or anticoagulant treatment, refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the affinity and specificity of binding of a positron emitter-labeled anti-Dimer antibody (64Copper) to fresh blood thrombus in vitro. | Day +0
  Evaluation of the binding rate of a 64Copper-labeled D-dimer-specific monoclonal antibody (64Cu-Antibody) on fresh blood thrombus from healthy donors. The rate of binding will be assessed by measuring the radioactivity present on the thrombus (64Cu-Antibody bound to the thrombus) and the radioactivity present in the supernatant (64Cu-Antibody not bound to the thrombus).

SECONDARY OUTCOMES:
Optimize the antibody concentration required for the most effective tracer binding (64Cu-Antibody) to the thrombus. | Day +0
  Determination of the optimum 64Cu-Antibody concentration for the most effective thrombus labeling. Incorporate increasing amounts of 64Cu Antibody concentration, and measure the amount of binding to fresh thrombus and to the supernatant.

CONTACTS AND LOCATIONS:
Locations (1):
- Etablissement francais du sang, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided